CLINICAL TRIAL: NCT06622486
Title: First-in-human Phase 1/2 Trial of EGL-001 in Adult Patients with Selected Advanced And/or Metastatic Solid Tumors
Brief Title: First-in-human Trial of EGL-001 in Patients with Selected Advanced And/or Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Egle Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: EGL-121; 2024-512921-10-00 (EU CTIS Number)
Record Dates: First submitted 2024-09-26; First posted 2024-10-02 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Solid Tumor, Adult

STUDY DESIGN:
Intervention Model Description: Dose escalation followed by combination therapy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (10):
- Monotherapy EGL-001 Dose Level 1 (Experimental): EGL-001 Dose Level 1
  Interventions: Drug: EGL-001
- Monotherapy EGL-001 Dose Level 2 (Experimental): EGL-001 Dose Level 2
  Interventions: Drug: EGL-001
- Monotherapy EGL-001 Dose Level 3 (Experimental): EGL-001 Dose Level 3
  Interventions: Drug: EGL-001
- Monotherapy EGL-001 Dose Level 4 (Experimental): EGL-001 Dose Level 4
  Interventions: Drug: EGL-001
- Monotherapy EGL-001 Dose Level 5 (Experimental): EGL-001 Dose Level 5
  Interventions: Drug: EGL-001
- Monotherapy EGL-001 Dose Level 6 (Experimental): EGL-001 Dose Level 6
  Interventions: Drug: EGL-001
- Monotherapy EGL-001 Dose Level 7 (Experimental): EGL-001 Dose Level 7
  Interventions: Drug: EGL-001
- Combination therapy with EGL-001 dose Level x (Experimental): EGL-001 Dose Level x in combination with anti-PDL1
  Interventions: Drug: EGL-001
- Combination therapy with EGL-001 dose Level y (Experimental): EGL-001 Dose Level y in combination with anti-PDL1
  Interventions: Drug: EGL-001
- Combination therapy with EGL-001 dose Level z (Experimental): EGL-001 Dose Level z in combination with anti-PDL1
  Interventions: Drug: EGL-001

INTERVENTIONS:
Drug: EGL-001 — IV administration

SUMMARY:
This multicenter, open-label, first-in-human, Phase 1/2 study consists of a Part 1 (Phase 1) open-label dose escalation of EGL-001 administered as a single agent and in combination with an anti-PD(L)-1 treatment, followed by a Part 2 (Phase 2) open-label dose expansion of EGL-001 administered at the RP2D in patients with recurrent and/or metastatic solid tumors as monotherapy and/or combination therapy with anti-PD(L)-1.

DETAILED DESCRIPTION:
In approximately 4 centers in France and 4 centers in Spain, 30 to 50 patients will be included in the dose escalation Part 1 of the trial. Number of participating countries and sites as well as patients will be defined based on Part 1 for Part 2 dose expansion phase.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent
2. Female or male patients, aged at least 18 years
3. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
4. Life expectancy of at least 3 months as assessed by the investigator
5. Patients with confirmed locally advanced, unresectable, or metastatic solid tumors who have been previously treated with SoC and are no longer eligible for other therapies
6. Patients who have been treated with an ICI treatment as monotherapy or in combination as SoC
7. Have recovered from previous treatment
8. At least 1 measurable lesion according to RECIST Version 1.1
9. Adequate hematological, hepatic, and renal functions
10. Negative blood pregnancy test at screening for women of childbearing potential
11. Highly effective contraception during the study period and for 6 months after the last study treatment administration for WOCBP, and for male patients who are sexually active with WOCBP. Highly effective contraception methods are defined as:

    * Hormonal methods of contraception including combined oral contraceptive pills, vaginal ring, injectable, implants, intrauterine devices such as Mirena and nonhormonal intrauterine devices such as ParaGard for WOCBP patients or male patients' WOCBP partners
    * Tubal ligation
    * Vasectomy

    In addition to highly effective contraception, participating male patients:
    * Must use a condom during the study period and for 3 months after the last study treatment administration when engaging in any activity that allows for exposure to ejaculate
    * Must refrain from donating sperm
12. Must agree to abstain from donating blood while taking study drug and for 3 months following discontinuation of study treatment
13. Able to understand the character and individual consequences of clinical trial

Exclusion Criteria:

1. Patients with central nervous system metastases and/or leptomeningeal carcinomatosis with some exceptions
2. Patients with active or a documented history of autoimmune disease, immune deficiency or syndrome that required systemic corticoids (except the allowed dose) or immunosuppressive medications
3. Patients who received a previous ICI like anti-PD(L)-1 or an agent directed to another stimulatory or co-inhibitory T-cell receptor and was discontinued from that treatment due to toxicity
4. Patients under chronic treatment with systemic corticosteroids or other immunosuppressive drugs for a period of at least 4 weeks and whose treatment was not stopped 2 weeks prior to the first study treatment, with exceptions. Steroids with no or minimal systemic effect (topical, inhalation) are allowed
5. Patients with history of or current interstitial lung disease or fibrosis, and patients with pneumonitis
6. Other active malignancy requiring active intervention
7. Patients with previous malignancies other than the target malignancy to be investigated in this trial, unless a complete remission was achieved and no additional therapy is required during the study period
8. Patient with any organ transplantation, including allogeneic stem cell transplantation
9. Known severe hypersensitivity reactions to monoclonal antibodies, any history of anaphylaxis, or uncontrolled asthma
10. Any known allergy or severe reaction to any component of anti-CTLA-4 or anti-PD(L)-1 drug product
11. Significant chronic or acute infections requiring systemic therapy including SARS-CoV-2 (COVID-19) PCR positive testing
12. Clinically significant active cardiovascular disease
13. Any other medical conditions or psychological disorders that would increase the safety risk to the patient or interfere with participation of the patient or the evaluation of the clinical study in the opinion of the investigator
14. Pregnant, breastfeeding, or expecting to conceive or father children within the projected duration of the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-09-27 (Actual); Primary Completion 2027-01-23 (Estimated); Study Completion 2027-01-23 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety, tolerability, dose-limiting toxicities (DLTs) and the maximum tolerated dose (MTD) leading to the recommended Phase 2 doses (RP2Ds) | Day 1 up to 90 days after last dose
  DLTs occurrence per dose level of EGL-001 during the DLT period (number)
To evaluate the safety, tolerability, dose-limiting toxicities (DLTs) and the maximum tolerated dose (MTD) leading to the recommended Phase 2 doses (RP2Ds) | Day 1 up to 90 days after last dose
  Proportion of patients with adverse events (AEs) (%)
To evaluate the safety, tolerability, dose-limiting toxicities (DLTs) and the maximum tolerated dose (MTD) leading to the recommended Phase 2 doses (RP2Ds) | Day 1 up to 90 days after last dose
  Proportion of patients with treatment-emergent AEs (TEAEs) (%)
To evaluate the safety, tolerability, dose-limiting toxicities (DLTs) and the maximum tolerated dose (MTD) leading to the recommended Phase 2 doses (RP2Ds) | Day 1 up to 90 days after last dose
  Proportion of patients with serious AEs (SAEs) (%)

SECONDARY OUTCOMES:
To evaluate the preliminary antitumor efficacy (according to RECIST v1.1) | From Dose 1 to to the date of first documented tumor progression or death due to any cause, whichever occurs first.
  ORR: the proportion of patients with complete response (CR) or partial response PR), based on local evaluations using RECIST Version 1.1. (%)
To evaluate the preliminary antitumor efficacy (according to RECIST v1.1) | From Dose 1 to to the date of first documented tumor progression or death due to any cause, whichever occurs first.
  Disease control rate (DCR): the proportion of patients with CR, PR, or stable disease (SD), and assessment of DCR at 6 months (%)
To evaluate the preliminary antitumor efficacy (according to RECIST v1.1) | From Dose 1 to to the date of first documented tumor progression or death due to any cause, whichever occurs first.
  Duration of overall response (DoR): applies only to patients with CR or PR. The start date is the date of first documented response (CR or PR), and the end date is the date of first documented disease progression or the date of death due to underlying cancer (months)
To evaluate the preliminary antitumor efficacy (according to RECIST v1.1) | From Dose 1 to to the date of first documented tumor progression or death due to any cause, whichever occurs first.
  PFS: time from the date of first study treatment administration to the date of first documented tumor progression or death due to any cause, whichever occurs first (months)
To evaluate the preliminary antitumor efficacy (according to RECIST v1.1) | From Dose 1 to to the date of first documented tumor progression or death due to any cause, whichever occurs first.
  OS: time from the date of first study treatment administration to the date of death due to any cause. If a patient is not known to have died at the cut-off date for analysis, survival will be censored at the date of last contact (months)

CONTACTS AND LOCATIONS:
Overall Officials: Pejvack Motlagh, MD, Study Director — Egle Therapeutics
Locations (8):
- France (4):
  - Centr Georges Francois Leclerc, Dijon
  - Institut Regional Du Cancer De Montpellier, Montpellier
  - Institut Curie, Paris
  - Institut Gustave Roussy, Paris
- Spain (4):
  - Hospital Universitari Vall D Hebron, Barcelona
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Clinica Universidad De Navarra, Pamplona
  - Hospital Clinico Universitario De Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No
Consequences (RA approval, data protection, operations for datamanagement, impact on IP, on budget…) for sharing IPD are not understood by Egle-Tx. This will be done at a later stage if necessary.